CLINICAL TRIAL: NCT04453852
Title: A Randomised, Controlled, Phase 1 Study to Evaluate the Safety and Immunogenicity of a Candidate Adjuvanted Recombinant Protein SARS-COV-2 Vaccine in Healthy Adult Subjects
Brief Title: Monovalent Recombinant COVID19 Vaccine
Acronym: COVAX19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxine Pty Ltd (Industry)
Collaborators: Central Adelaide Local Health Network Incorporated (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13110
Record Dates: First submitted 2020-06-03; First posted 2020-07-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus Infection; COVID
Keywords: COVID19; coronavirus; vaccine; adjuvant
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — COVID-19 Vaccines; SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomised controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Non-blind Staff administering vaccine do not participate in any other aspects of the study. Remaining trial staff and participant are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Spike antigen (25ug) + 15 mg Advax-2 adjuvant
  Interventions: Biological: COVID19 vaccine
- Group B (Placebo Comparator): Saline
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: COVID19 vaccine — COVID19 recombinant spike protein with Advax-SM adjuvant
  Other Names: COVAX-19 vaccine
  Arms: Group A
Biological: Saline — Saline control
  Other Names: Saline control
  Arms: Group B

SUMMARY:
This is a study to test a new vaccine (Covax-19) against COVID-19. COVID-19 is a potentially deadly disease that is caused by a new strain of coronavirus called SARS-CoV-2. To date, SARS-CoV-2 has infected over 4 million people worldwide resulted in the deaths of over three hundred thousand people.

DETAILED DESCRIPTION:
Human infections with zoonotic coronaviruses including severe acute respiratory syndrome coronavirus (SARS CoV), Middle East respiratory syndrome-associated coronavirus (MERS CoV) and now 2019 SARS-CoV-2, all pose major human public health threats with high case fatality rates. The outbreak of SARS-CoV-2, which shares high similarity with SARS-CoV in its viral genome, has so far caused more than 4,736,000 cases worldwide (as of May 17, 2020) with 3131,545 deaths, resulting in an estimated overall mortality rate of 4-5%. It has a particularly high mortality rate in elderly people and those with chronic disease. To fight the current outbreak and prepare for future human outbreaks of similar coronaviruses, development of a safe and effective SARS-COV-2 vaccine remains a high priority. The fatality rate in the elderly is very high, being 8% for those over 70 and over 20% for those over 80. Notably, over 16% of the Australian population is aged 65 or older. Currently there is no way to control infection with SARS-COV-2 other than minimise exposure by social isolation.

Development of a vaccine against COVID-19 would deliver major public health and economic benefits for Australia, with potential to prevent numerous deaths, particularly among the Australian elderly, reducing the burden on hospital ICUs, helping to alleviate public concern, and ultimately allowing the Australian economy to return as fast as possible to normal.

SARS-CoV and SARS-CoV-2 are both closely related enveloped, single positive-stranded RNA viruses, with one genome encoding a non-structural replicase polyprotein and structural proteins, including spike (S), envelope (E), membrane (M) and nucleocapsid (N) proteins. SARS virus neutralizing antibodies were shown to be directed against the S protein. S protein can be cleaved into S1 and S2 subunits by proteases and within the S1 subunit there is a receptor-binding domain (RBD), which was shown to bind angiotensin-converting enzyme 2 (ACE2), which mediates SARS virus entry into cells. SARS-CoV-2 spike protein similarly binds ACE2 for cellular entry. Hence a recombinant SARS-CoV-2 spike protein vaccine that induces neutralising antibody against the virus should be effective against SARS-CoV-2 infection just as seen for SARS CoV.

SARS-COV-2 vaccine design is best informed by previous experience with closely related SARS CoV vaccines. Antibodies against the coronavirus spike protein blocks infection. When recombinant SARS spike protein vaccines produced in insect cells were formulated with Advax adjuvant, this enhances neutralizing antibody and T cell responses which translate into rapid lung viral clearance. Based on experience with developing successful and safe SARS and MERS vaccines, Covax-19 vaccine design is based on recombinant insect cell- expressed SARS-COV-2 spike protein formulated with Advax-SM adjuvant. The vaccine is based on recombinant expression of the ecto-domain of spike protein in insect cells. Insect cell expression of recombinant protein is a well characterised platform, allowing standardised procedures to be rapidly transferred to other facilities around the world. In response to the 2009 H1N1 influenza pandemic, roll-out of a pandemic vaccine based on hemagglutinin protein was extremely fast, with the first cGMP batches of vaccine produced within 6 weeks of virus discovery, and the first human trial subject dosed at Flinders just under 3 months after virus discovery . The use of Advax adjuvant doubled the seroconversion and seroprotection rates while maintaining vaccine tolerability and safety. Recombinant proteins manufactured using this method and formulated with Advax adjuvants have been found to be effective and safe in multiple human trials, including of H1N1/2009 and H5N1 (NCT02335164) and H7N9 (NCT03038776) influenza vaccines.

Covax-19 consists of highly purified recombinant SARS-COV-2 spike protein plus Advax-SM adjuvant in a sterile solution for intramuscular injection. COVAX-19™ vaccine is manufactured using a Sf9 platform. Advax-CpG adjuvant has previously been well tolerated and effective in trials of hepatitis B, H5N1 (NCT02335164) and H7N9 (NCT03038776) influenza vaccines and has recently been tested by the NIH in a US multicentre clinical trial with 2 quadrivalent seasonal influenza vaccines (NCT03945825).

COVAX-19™ vaccine is designed to elicit an immune response against SARS-CoV-2 with generation of neutralising antibodies against its spike protein that prevent the virus attaching to the human ACE2 receptor in the respiratory epithelium. It is also designed to induce T cells against the spike protein.

Study hypotheses

* COVAX-19 vaccine is safe and well tolerated in adult human subjects
* COVAX-19 vaccine will induce durable high titer neutralising antibodies and T cell responses against SARS-COV-2 virus.

ELIGIBILITY:
Inclusion criteria

* Subjects eligible to participate in this trial had to meet all of the following inclusion criteria:
* Provide written informed consent prior to initiation of any study procedures.
* Healthy males or non-pregnant females, aged 18 years to 65 years inclusive.
* Women of childbearing potential2 must use an acceptable contraception method3 from at least 30 days before study vaccination until 90 days after study vaccination.

  2Not sterilized via, bilateral oophorectomy, salpingectomy, hysterectomy, (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal.

  3Includes full abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more barrier methods such as condoms, effective intrauterine devices, tubal ligation, and approved hormonal methods such as implants, injectables or oral contraceptives ("the pill").
* Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination
* Are able to understand and comply with planned study procedures and be available for all study visits.

Exclusion criteria

* • Have an acute illness, as determined by the site Principal Investigator (PI) or appropriate sub-investigator, within 72 hours prior to study vaccination.
* Have a history of documented COVID-19 infection or a known positive COVID-19 antibody test.
* Liver function tests (ALT, AST or GGT) > 2 times upper limit of normal
* eGFR <55 mL/min/1.73 m2
* Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
* Use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to study vaccination.
* Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy.
* Have known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection.
* Have a history of severe systemic reactions following previous immunization with licensed or unlicensed vaccines.
* Have a history of Guillain-Barré Syndrome.
* Have known hypersensitivity or allergy to insect stings or other components of the study vaccine.
* Have a history of epilepsy or febrile convulsions
* Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).
* Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
* Have any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations as determined by the site PI or appropriate sub-investigator.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 5 years prior to study vaccination.
* Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
* Have taken high-dose inhaled corticosteroids within 30 days prior to study vaccination.
* Female participants who are breastfeeding or plan to breastfeed from the time of the first study vaccination through 30 days after the last study vaccination.
* Positive urine or serum pregnancy test within 24 hours prior to any study vaccination
* Received an experimental agent within 30 days prior to the study vaccination or expect to receive another experimental agent during the trial-reporting period.
* Have any medical disease or condition that, in the opinion of the Investigator, is a contraindication to study participation.
* Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation. *Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
* Any participant whose enrolment, in the opinion of the investigator, would be detrimental to the participant or the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 1 week post immunisation
  Incidence of Adverse Events 1 week post immunisation
COVID19 antibody titers | 3 weeks post second immunisation
  COVID19 antibody titers post immunisation
COVID19 T cell immunogenicity | 3 weeks post second immunisation
  Frequency of COVID19 spike specific T cells 1-3 weeks post second immunisation

CONTACTS AND LOCATIONS:
Overall Officials: David Gordon, MBBS, Ph.D, Principal Investigator — CALHN
Locations (1):
- PARC,, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No